CLINICAL TRIAL: NCT02170987
Title: Assessment of Electrophysiological Effects of 150 mg and 600 mg of Dabigatran Etexilate as Single Dose on the QT Interval in Healthy Female and Male Subjects. A Randomised, Placebo Controlled, Double-blind Three-way Crossover Study With an Open Label Positive Control (Moxifloxacin)
Brief Title: Assessment of Electrophysiological Effects of Dabigatran Etexilate as Single Dose on the QT Interval in Healthy Female and Male Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1160.54
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Moxifloxacin

ARMS (4):
- Dabigatran etexilate low (Experimental)
  Interventions: Drug: Dabigatran etexilate low
- Dabigatran etexilate high (Experimental)
  Interventions: Drug: Dabigatran etexilate high
- Placebo to dabigatran etexilate (Placebo Comparator)
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Dabigatran etexilate low
  Arms: Dabigatran etexilate low
Drug: Dabigatran etexilate high
  Arms: Dabigatran etexilate high
Drug: Moxifloxacin
  Arms: Moxifloxacin
Drug: Placebo
  Arms: Placebo to dabigatran etexilate

SUMMARY:
To investigate if dabigatran has a clinically relevant impact on the cardiac electrophysiology that is manifest as prolongation in QT-interval.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female (at least 1/3) and male (at least 1/3) volunteers as determined by the results of screening according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, HR), 12-lead ECG, clinical laboratory tests
2. Age >= 18 and Age <= 65 years
3. BMI >= 20.0 and BMI <=29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including BP, pulse rate (PR) and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
8. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
10. Participation in another trial with an investigational drug within two months prior to administration or during the trial
11. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
12. Inability to refrain from smoking on trial days
13. Alcohol abuse (more than 60 g/day)
14. Drug abuse
15. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
16. History of any bleeding disorder or acute blood coagulation defect
17. Hypersensitivity to moxifloxacin and/or related drugs of this class
18. Excessive physical activities (within one week prior to administration or during the trial)
19. Any laboratory value outside the reference range that is of clinical relevance
20. Inability to comply with dietary regimen of study centre
21. History of additional risk factors for Torsade des Pointes (e.g. heart failure, hypokalemia, family history of long QT syndrome)
22. Any screening ECG value outside of the reference range of clinical relevance including, but not limited to heart rate of >80 bpm or <45 bpm, PR interval >220 ms, QRS interval >120 ms, QT interval >470 ms or QTcB or QTcF >450 ms

    For female subjects:
23. Pregnancy
24. Positive pregnancy test
25. No adequate contraception e.g. oral contraceptives, sterilisation, intrauterine device (IUD)
26. Inability to maintain this adequate contraception during the whole study period
27. Lactation period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-03; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean time-matched QTc Interval | at 1.5, 2, and 3 hours following administration

SECONDARY OUTCOMES:
Mean of the QTcI values of all ECGs | from 1 to 6 hours following administration
Change from baseline of the QTcI | from 1 to 24 hours following administration